CLINICAL TRIAL: NCT04022473
Title: A Randomized, Double-Blind Study to Compare Gastrointestinal Tolerability Following Oral Administration of Bafiertam™ (Monomethyl Fumarate) or Tecfidera® (Dimethyl Fumarate) to Healthy Male and Female Volunteers
Brief Title: Study to Compare GI Tolerability Following Oral Administration of Bafiertam™ or Tecfidera to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Banner Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLS-11-109
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
Keywords: Gastrointestinal
MeSH Terms: conditions — Multiple Sclerosis | interventions — monomethyl fumarate; Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bafiertam (Experimental): oral capsules administered twice daily
  Interventions: Drug: Bafiertam
- Tecfidera (Active Comparator): oral capsules administered twice daily
  Interventions: Drug: Tecfidera

INTERVENTIONS:
Drug: Bafiertam — Over-encapsulated capsule to mask treatment
  Other Names: monomethyl fumarate
  Arms: Bafiertam
Drug: Tecfidera — Over-encapsulated capsule to mask treatment
  Other Names: dimethyl fumarate
  Arms: Tecfidera

SUMMARY:
The primary objective of the study is to compare in healthy subjects, the GI tolerability of bioequivalent doses of Bafiertam™(monomethyl fumarate) and its pro-drug Tecfidera® (dimethyl fumarate).

Secondary objective of this study is to compare the safety and tolerability of Bafiertam™ and Tecfidera® when administered orally following bioequivalent dose regimens in healthy subjects.

DETAILED DESCRIPTION:
Subjects randomized (1:1) to either Bafiertam (monomethyl fumarate) or Tecfidera (dimethyl fumarate) will enter a double-blind titration period where they will receive either Bafiertam 95 mg twice daily (BID) or Tecfidera 120 mg BID for 7 days. Following the titration period, they will enter a maintenance period in which they will receive Bafiertam 190 mg BID or Tecfidera 240 mg BID for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females.
2. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
3. Body Mass Index within 18.0 - 34.0 kg/m2, inclusive

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic, renal/genitourinary, Gastrointestinal (GI), cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
2. Clinically significant history or presence of any clinically significant GI pathology unresolved GI symptoms, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first study drug administration, as determined by the PI/Sub-Investigator.
3. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
4. Subject with abnormal baseline laboratory values deemed to be clinically significant by the Investigator.
5. Lymphocyte count <1.5x 10^9/L.
6. Known history or presence of: Alcohol abuse or dependence within one year prior to first study drug administration; Drug abuse or dependence; Hypersensitivity or idiosyncratic reaction to DMF, its excipients, and/or related substances; Progressive multifocal leukoencephalopathy (PML); Fanconi syndrome; Flushing (e.g., warmth, redness, itching, and burning sensation); Low white blood cell count (lymphopenia);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) in each of the individual symptoms over the treatment period. | 5 weeks
  The symptoms measured are (1) nausea, (2) vomiting, (3) diarrhea, (4) upper abdominal pain, (5) lower abdominal pain, (6) constipation, (7) bloating, and (8) flatulence

SECONDARY OUTCOMES:
Comparison of the Modified Overall Gastrointestinal Symptom Scale (MOGISS) composite score | 5 weeks
  The MOGISS assesses global GI events (defined as one or more of the following symptoms: nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, constipation, bloating, and flatulence) and their effect on the patient during the 24 hours before each morning dose. The events items are rated on a 10-point numerical rating scale, where 0 = no events, 1 to 3 = mild events, 4 to 6 = moderate events, 7 to 9 = severe events, and 10 = extreme events. The MOGISS Total (sum of 8 scores) range is 0 (no symptoms) to 80 (worst possible symptoms) and the MOGISS Composite (average of 8 scores) range is 0 (no symptoms) - 10 (worst possible symptoms).
The number of days that a subject experiences at least one GI symptom. | 5 weeks
  Number of days with at (as reported on the MOGISS) with a severity score of at least 1
AUC in the MOGISS total score within in each subject over the treatment period | 5 weeks
  Defined as the daily total of all 8 individual symptom scores within each subject
Frequency, severity, and duration of overall GI events using the MOGISS. | 5 weeks
  Frequency, severity and duration of overall GI events will be completed using the MOGISS for each week of study treatment as well as for the overall study treatment period.
Safety and tolerability outcomes: incidence rates of all non GI-adverse events | 5 weeks
  Subject incidence rates of all non GI-adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Doisy, MD, Principal Investigator — BioPharma Services Inc.
Locations (1):
- BioPharma Services, Inc., Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentiﬁcation (text, tables, ﬁgures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 12 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identiﬁed for this purpose.
  The stated purpose of the analysis as to be for individual participant data meta-analysis.